CLINICAL TRIAL: NCT05609955
Title: Effects Of Additional MgSO4 30 Mg/KgBW Intravenous and Ketorolac : Study to Assess Pain And Opioid Consumption in Post Lower Extremity Orthopedic Surgery
Brief Title: Effects Of Additional MgSO4 30 Mg/KgBW Intravenous and Ketorolac
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, PhD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUAnes124
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia; Pain, Postoperative; Surgery; Opioid Use
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MgSO4 (Experimental): The treatment group received intravenous magnesium sulfate therapy with a 20% magnesium sulfate regimen, 39mg/kg body weight dissolved in 100ml NaCl in 1 hour intravenously.
  Interventions: Drug: MgSO4
- Placebo (Placebo Comparator): The treatment group who received intravenous placebo therapy with a regimen of 100 ml NaCl in 1 hour intravenous
  Interventions: Drug: MgSO4

INTERVENTIONS:
Drug: MgSO4 — The treatment group who received intravenous magnesium sulfate therapy with 20% magnesium sulfate regimen, 30mg/kg body weight dissolved in 100ml NaCl in 1 hour intravenously

SUMMARY:
This study aims to compare two groups of post-orthopedic patients who received a standard regimen, namely ketorolac 30mg, to the second group, which was given the standard regimen and adjuvant magnesium sulfate 30mg/kgBW 1 hour preoperatively. If it is proven useful, it is hoped that pain will be more controlled, reduce pain complications, reduce treatment costs, and reduce the duration of hospital stays.

DETAILED DESCRIPTION:
The study design used was a randomized controlled trial (RCT) with double blinds. Double blind because neither the patient, the lead investigator, nor the investigator on record knew the drug or placebo that was administered. Research subjects were selected consecutively in patients who will undergo lower extremity surgery at the Cipto Mangunkusumo National Central General Hospital. Forty-eight research subjects will be divided into two groups, namely the group given Intravenous Magnesium Sulfate 30 mg/kgBW and the group given a placebo. Research subjects were randomized by type of surgery using randomization software by research assistants. The results of randomization were not known to the patient, the principal investigator, or the researcher taking notes.

This study aims to determine the effect of adding 30 mg/kg body weight of intravenous MgSO4 to 30 mg of ketorolac on the degree of pain and the need for opioids after lower extremity surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lower extremity orthopedic surgery under general anaesthesia.
* Patients aged 18-60 years.
* Physical status ASA 1-3
* Willing to participate in research.

Exclusion Criteria:

* Patients who are hemodynamically unstable.
* Patients with decreased renal function
* Patients with skeletal muscle disorders.
* Patients with Ketorolac allergy
* Patients with morphine allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 24 hour
  The scale for measuring pain felt by the patient is in the form of a horizontal straight line 100 mm long. In the VAS examination, the patient is asked to point to a point along the line that reflects the degree of pain felt. There is a millimeter ruler for calculating the VAS score. A score of 0 = no pain and a score of 10 = unbearable severe pain.

SECONDARY OUTCOMES:
Morphine consumption | 24 hour
  The number of milligrams (mg) of intravenous morphine in the first 24 hours postoperatively using a PCA device.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No